CLINICAL TRIAL: NCT06508502
Title: Pancreatitis - Microbiome as Predictor of Severity II
Acronym: P-MAPS II
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Christoph Ammer-Herrmenau, Dr., University Medical Center Goettingen
Other Study IDs: 2024-03261
Record Dates: First submitted 2024-07-10; First posted 2024-07-18 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Acute Pancreatitis; Acute Pancreatitis With Infected Necrosis
Keywords: Pancreatitis; Microbiome
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal and rectal swabs Stool Plasma All samples are stored at -80°C within 30 minutes after collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Revised Atlanta classifiaction (RAC) I - mild: No local or systemic complication
- Revised Atlanta classifiaction (RAC) II - moderate severe: Local complications as necrosis or fluid collection or organ failure < 48h
- Revised Atlanta classifiaction (RAC) III - severe: Organ failure > 48h

SUMMARY:
The goal of this observational study is to evaluate the orointestinal microbiome and microbial derived metabolome in patients suffering from acute pancreatitis as a biomarker for severity. The main questions it aims to answer are:

* Can the orointestinal microbiome robustly predict the course of acute pancreatitis?
* How does the microbiome impact the severity of an acute pancreatitis?

Buccal/ rectal swabs, plasma and stool is collected from patients with acute pancreatitis within 48h after hospital admission.

DETAILED DESCRIPTION:
Despite intensive research, early prediction of the course of acute pancreatitis (AP) is still not satisfactorily possible. Results of a European multicenter study showed that the intestinal microbiome is superior to established scores as a marker of severity in patients with AP. Hereby, a classifier was established using 16 differentially abundant rectal species and systemic inflammatory response syndrome (SIRS) and achieved an AUROC of 85%. Surprisingly, all species in the severe AP group were members of taxonomic families known for their short-chain fatty acid (SFCA) production. This observation contrasts with translational pancreatitis studies in mice. Based on these publications, a clinical trial is currently being initiated to treat severe AP with SCFA (NCT06147635). However, previous well-designed RCT that analyzed the effects of probiotics in predicted severe AP resulted in a worse outcome for patients in the probiotic arm. Consequently, national and international guidelines recommend against the usage of probiotics in AP.

Collectively, more research is needed to further elucidate the role of the oro-intestinal microbiota in the development of severe AP. To validate the results of previously mentioned multicenter study and to profoundly analyze the role of microbial metabolites and the fungeome, patients with AP will be prospectively recruited.

1. Buccal and rectal swabs, stool and plasma will be obtained to analyze the orointestinal microbiome and microbial derived metabolites.
2. Centers from different continents with different ethical background and dietary habits will enroll patients to gain a more generalizable microbial profile.
3. Microbial shifts were observed between severe AP (RAC 3) and mild/ moderate severe (RAC 1+2).
4. It is expected that the microbial compositions change during the inflammatory process upon early phase of pancreatitis. To minimize this microbial alternating effect a short time frame from hospital admission to recruitment (48h) is set.

ELIGIBILITY:
Inclusion Criteria:

* Patients with initial diagnosis (< 48h) of acute pancreatitis
* Age ≥ 18 years
* Patients able to understand/ give their written consent

Exclusion Criteria:

* Recurrent acute pancreatitis (>2 previous episodes)
* Clinical or imaging signs of chronic pancreatitis
* Referred patients with length of hospital stay > 48h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute pancreatitis within 48h after hospital admission. Acute pancreatitis is defined if 2 of the following criteria are fullfilled.
  1. Lipase > 3x the upper limit
  2. Typical abdominal pain (belt-like upper abdominal pain)
  3. Characteristic CT findings
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Novel microbiome species and/or functional metabolic pathways that are associated with the severity of acute pancreatitis | until discharge (up to 90 days)
  To assess the microbial diversity and differential abundances of species within buccal and rectal swabs analyzed by ONT sequencing followed by prediction of metabolic pathways and metabolites using tools such as Megan6 and GapSeq stratified by the Revised Atlanta Classification and severity (necrotic collections that require intervention and/or organ failure >48h), adjusted for multiple individual confounders.
Classifier developed based on differentially regulated metabolites | Until discharge (up to 90 days)
  To assess the metabolite (predicted in 1. Primary endpoint) levels in stool and plasma samples by targeted metabolomics to develop a classifier based on differentially regulated metabolites to assess its discriminatory power in predicting Revised Atlanta Classification and severity.

SECONDARY OUTCOMES:
Mortality | up to 1096 days (3 years)
  Association of mortality with microbial diversity and differential abundance and differentially regulated metabolites adjusted for multiple individual confounder. Long-term outcomes will be assessed in the current cohort (P-MAPS II), as well as in the previously established P-MAPS I cohort (NCT04777812).
Length of hospital stay | up to 90 days
  Association of length of hospital stay with microbial diversity and differential abundance and differentially regulated metabolites adjusted for multiple individual confounder.
Post-discharge exocrine and endocrine insufficiency | up to 90 days
  Association of post-discharge exocrine and endocrine insufficiency with microbial diversity and differential abundance and differentially regulated metabolites adjusted for multiple individual confounder. Long-term outcomes will be assessed in the current cohort (P-MAPS II), as well as in the previously established P-MAPS I cohort (NCT04777812).
Post-discharge re-intervention | up to 1096 days (3 years)
  Association of post-discharge re-intervention with microbial diversity and differential abundance and differentially regulated metabolites adjusted for multiple individual confounder. Long-term outcomes will be assessed in the current cohort (P-MAPS II), as well as in the previously established P-MAPS I cohort (NCT04777812).
Recurrent/chronic pancreatitis rate | up to 1096 days (3 years)
  Association of recurrent/chronic pancreatitis rate with microbial diversity and differential abundance and differentially regulated metabolites adjusted for multiple individual confounder. Long-term outcomes will be assessed in the current cohort (P-MAPS II), as well as in the previously established P-MAPS I cohort (NCT04777812).
Volatile organic compounds | Until discharge (up to 90 days)
  Assessment of volatile organic compounds (VOCs) in a subset of the study cohort (n = 60), including group comparisons based on the revised Atlanta classification and severity, as well as correlation of VOC concentrations with corresponding plasma levels.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Goettingen, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Capurso G, Ponz de Leon Pisani R, Lauri G, Archibugi L, Hegyi P, Papachristou GI, Pandanaboyana S, Maisonneuve P, Arcidiacono PG, de-Madaria E. Clinical usefulness of scoring systems to predict severe acute pancreatitis: A systematic review and meta-analysis with pre and post-test probability assessment. United European Gastroenterol J. 2023 Nov;11(9):825-836. doi: 10.1002/ueg2.12464. Epub 2023 Sep 27. PMID 37755341
- [Background] Ammer-Herrmenau C, Antweiler KL, Asendorf T, Beyer G, Buchholz SM, Cameron S, Capurso G, Damm M, Dang L, Frost F, Gomes A, Hamm J, Henker R, Hoffmeister A, Meinhardt C, Nawacki L, Nunes V, Panyko A, Pardo C, Phillip V, Pukitis A, Rasch S, Riekstina D, Rinja E, Ruiz-Rebollo ML, Sirtl S, Weingarten M, Sandru V, Woitalla J, Ellenrieder V, Neesse A. Gut microbiota predicts severity and reveals novel metabolic signatures in acute pancreatitis. Gut. 2024 Feb 23;73(3):485-495. doi: 10.1136/gutjnl-2023-330987. PMID 38129103
- [Background] Ammer-Herrmenau C, Neesse A. Response to: short-chain fatty acids in patients with severe acute pancreatitis: friend or foe? Gut. 2024 Nov 11;73(12):e39. doi: 10.1136/gutjnl-2024-332236. No abstract available. PMID 38453356
- [Background] van den Berg FF, Besselink MG, van Santvoort H. Short-chain fatty acids in patients with severe acute pancreatitis: friend or foe? Gut. 2024 Nov 11;73(12):e34. doi: 10.1136/gutjnl-2024-332129. No abstract available. PMID 38360070
- [Background] Besselink MG, van Santvoort HC, Buskens E, Boermeester MA, van Goor H, Timmerman HM, Nieuwenhuijs VB, Bollen TL, van Ramshorst B, Witteman BJ, Rosman C, Ploeg RJ, Brink MA, Schaapherder AF, Dejong CH, Wahab PJ, van Laarhoven CJ, van der Harst E, van Eijck CH, Cuesta MA, Akkermans LM, Gooszen HG; Dutch Acute Pancreatitis Study Group. Probiotic prophylaxis in predicted severe acute pancreatitis: a randomised, double-blind, placebo-controlled trial. Lancet. 2008 Feb 23;371(9613):651-659. doi: 10.1016/S0140-6736(08)60207-X. Epub 2008 Feb 14. PMID 18279948
- [Background] Beyer G, Hoffmeister A, Michl P, Gress TM, Huber W, Algul H, Neesse A, Meining A, Seufferlein TW, Rosendahl J, Kahl S, Keller J, Werner J, Friess H, Bufler P, Lohr MJ, Schneider A, Lynen Jansen P, Esposito I, Grenacher L, Mossner J, Lerch MM, Mayerle J; Collaborators:. S3-Leitlinie Pankreatitis - Leitlinie der Deutschen Gesellschaft fur Gastroenterologie, Verdauungs- und Stoffwechselkrankheiten (DGVS) - September 2021 - AWMF Registernummer 021-003. Z Gastroenterol. 2022 Mar;60(3):419-521. doi: 10.1055/a-1735-3864. Epub 2022 Mar 9. No abstract available. German. PMID 35263785
- [Background] Tenner S, Baillie J, DeWitt J, Vege SS; American College of Gastroenterology. American College of Gastroenterology guideline: management of acute pancreatitis. Am J Gastroenterol. 2013 Sep;108(9):1400-15; 1416. doi: 10.1038/ajg.2013.218. Epub 2013 Jul 30. PMID 23896955